CLINICAL TRIAL: NCT01407380
Title: A Phase 1, Open-Label, Dose-Escalation Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of Orally Administered PWT33597 Mesylate in Subjects With Advanced Malignancies
Brief Title: Study of PWT33597 Mesylate in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pathway Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PWT33597-101
Record Dates: First submitted 2011-07-21; First posted 2011-08-02 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Malignancies
Keywords: Advanced malignancies; solid tumors; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PWT33597 mesylate — PWT33597 taken orally daily for 28 consecutive days in 28 day cycle

SUMMARY:
This is a Phase 1 study evaluating the safety, pharmacokinetics, pharmacodynamics, and clinical effects of orally administered PWT33597 mesylate in subjects with advanced malignancies.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, dose-escalation study, to be conducted in 2 phases. The Dose Escalation Phase (up to 36 patients) will determine the MTD of PWT33597 mesylate and evaluate its safety and tolerability, PK, PD, and preliminary clinical effects; the subsequent Dose Confirmation Phase (up to 36 patients) will be a cohort expansion at or below the MTD of PWT33597 mesylate. Subjects will be treated with once-daily oral doses of PWT33597 in consecutive, 28-day cycles. Subjects will be evaluated regularly for safety. Subjects will return for a follow-up visit 28 days after completion of the last dose of study drug. Subjects who tolerate the drug and who do not experience progressive disease may continue to receive PWT33597 mesylate at the discretion of the principal investigator for up to 24 cycles

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. Pathologically confirmed advanced solid tumor or malignant lymphoma for which standard therapy proven to provide clinical benefit does not exist or is no longer effective.
3. Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤1
4. Evaluable disease, either measurable on physical examination or imaging by Response Evaluation Criteria in Solid Tumors (RECIST v1.1), or by the criteria of the International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma, or by informative tumor marker(s).
5. Laboratory values at screening:

   * Absolute neutrophil count ≥1,500 /mm3;
   * Platelets ≥100,000/mm3;
   * Total bilirubin ≤1.5 × the upper limit of normal (ULN);
   * AST (SGOT) ≤2.5 × the ULN;
   * ALT (SGPT) ≤2.5 × the ULN;
   * Serum creatinine ≤1.5 mg/dL or a measured creatinine clearance ≥60 mL/min; and
   * Negative serum beta-hCG test in women of childbearing potential (defined as women ≤50 years of age or history of amenorrhea for ≤12 months prior to study entry).
6. Patients with primary liver cancer or hepatic metastasis are eligible to enroll, provided that, at screening, the following criteria are met:

   * Total bilirubin is no higher than the ULN;
   * AST and ALT are each ≤5 × the ULN;
   * Severe liver dysfunction (Child-Pugh Class B or C) is not present; and
   * Patients with a history of esophageal bleeding have varices that have been sclerosed or banded and no bleeding episodes have occurred during the prior 6 months.
7. If there is a history of brain metastases treated with radiation therapy, the radiation therapy must have occurred at least 6 weeks prior to enrolment and the metastatic disease must have been stable since completion.
8. Willing and able to provide written Informed Consent and comply with the requirements of the study.
9. In addition, subjects enrolled in the Dose Confirmation Phase must meet the following criteria:

   * For subjects with solid tumors, measurable disease, using RECIST v1.1;
   * For subjects with malignant lymphoma, at least 1 lesion clearly measurable and >1.5cm transverse diameter in 2 perpendicular dimensions, per the criteria for International Working Group Revised Response Criteria for Malignant Lymphoma;
   * No prior treatment with an investigational PI3K, PI3K/mTOR, AKT or mTORC1/mTORC2 inhibitor (prior treatment with temsirolimus, everolimus, or ridaforolimus is allowed);
   * For subjects with colorectal cancer, evidence of lack of mutation in KRAS and BRAF, unless otherwise approved by the sponsor.
   * Tissue block or biopsy confirmation of PI3K alpha mutation on tumor genotyping.
   * Tumor accessible for pre- and post-treatment biopsy or cytology (in a subset of at least 5 subjects in each specific tumor type).

Exclusion Criteria:

1. Any chemotherapy, immunomodulatory drug therapy, anti-neoplastic hormonal therapy, immunosuppressive therapy, corticosteroids > 20 mg/day prednisone or equivalent (unless administered to prevent contrast material reactions during radiographic procedures), or growth factor treatment (eg, erythropoietin) within 14 days prior to initiation of study drug.
2. Presence of an acute or chronic toxicity of prior chemotherapy, with the exception of alopecia or peripheral neuropathy, that has not resolved to ≤ Grade 1, as determined by National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) v 4.0
3. Receipt of more than 5 prior regimens of cytotoxic chemotherapy unless prior approval is granted by the sponsor.
4. Radiotherapy within 4 weeks prior to baseline.
5. Receipt of radiotherapy to >25 % of bone marrow.
6. History of stem cell allotransplantation.
7. Major surgery within 28 days prior to initiation of study drug.
8. Life expectancy <12 weeks.
9. Active infection requiring systemic therapy.
10. Insulin-requiring diabetes mellitus, or presence of persistent fasting blood glucose >160 mg/dL.
11. Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
12. Known active hepatitis B or C or other active liver disease (other than malignancy).
13. Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
14. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to > 450 msec for males or > 470 msec for females.
15. Previous malignancy, except for non-basal-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, unless the tumor was treated with curative intent more than 2 years prior to study entry.
16. Concomitant treatment with, or anticipated use of, pharmaceutical or herbal agents which are potent inhibitors or inducers of cytochrome P450 3A4 enzymes, unless approved by the sponsor.
17. Use of any investigational agents within 4 weeks of baseline.
18. Pregnant or lactating female.
19. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the Principal Investigator, are effective and adequate for that patient's circumstances while on study drug and for 3 months afterward.
20. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (ie, a condom, with female partner using oral, injectable, or barrier method) while on study drug and for 3 months afterward.
21. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 2 years

SECONDARY OUTCOMES:
Number of patients whose tumor show objective response or stable disease by standard criteria | 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Pinnacle Hematology Oncology, Scottsdale, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee